CLINICAL TRIAL: NCT01233193
Title: Pharmacist Intervention Effect on the Medication Adherence and Blood Pressure Control in Treated Patients
Brief Title: The Effect of Pharmacist Intervention on Blood Pressure Control
Acronym: AFenPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: María José Faus Dáder, Pharmaceutical Care Research Group of the University of Granada
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DMM01-FAR-10
Record Dates: First submitted 2010-10-29; First posted 2010-11-03 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2010-02

CONDITIONS: Hypertension
Keywords: Home blood pressure measurement; Pharmaceutical Services; Medication adherence; hypertension management; Blood Pressure
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention group receive an pharmacist intervention (health education, Home Blood Pressure Monitoring and Referral to physician as needed) This group will be followed for 6 months
  Interventions: Behavioral: Health education, Home blood pressure monitoring
- Control (No Intervention): The control group receive usual care in the community pharmacy

INTERVENTIONS:
Behavioral: Health education, Home blood pressure monitoring — Health education (on hypertension, smoking, healthy diet, obesity, physical inactivity and adherence to antihypertensive medications and home blood pressure monitoring) . The patient will be referred to physician when needed. The patient will be followed up during 6 months.
  Other Names: pharmaceutical health education
  Arms: Intervention

SUMMARY:
The purpose of the study is to test if a Pharmacist Intervention Program with home blood pressure monitoring (HBPM) improves or controls pharmacological adherence and blood pressure levels in hypertensive patients under pharmacological treatment, compared to those who receive usual care in a community pharmacy setting.

DETAILED DESCRIPTION:
Hypertension is a major health concern worldwide due to its deleterious impact on the population in terms of excessive morbidity and mortality, especially when there is insufficient hypertension control and prevention at the community level.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders between the ages of 18 and 80 years, who access the pharmacy to fill their own prescription for hypertension.

Exclusion criteria:

* Patient living with an other Hypertensive patient treated with the same medications
* Pregnant women
* Hypertensive patients with levels of systolic/diastolic blood pressure ≥ 180mmHg/110mmHg
* Patient with secondary hypertension, kidney or liver failure
* Patients already included in a care program for hypertensive patients
* Patients with a new treatment for hypertension (less than 1 month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
blood pressure control | At 6 months
  Percentage of patients with controlled hypertension

SECONDARY OUTCOMES:
Adherence | At 6 months
  Percentage of adherent patients after 6 months within the trial

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jose Faus, PhD, Study Director — Universidad de Granada
Locations (2):
- Spain (2):
  - Community Pharmacies, Granada, Andalusia
  - Community Pharmacies, Jaén, Andalusia